CLINICAL TRIAL: NCT04325347
Title: Reducing Awakenings and Increasing Sleep Efficiency With Virtual Reality in Patients Suffering From Diabetic Polyneuropathy
Brief Title: VR in Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESOLVE
Record Dates: First submitted 2020-03-16; First posted 2020-03-27 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Virtual Reality will be provided to all participants, just before sleeping.
  Interventions: Other: Virtual Reality application
- Control (No Intervention): No specific intervention will be provided.

INTERVENTIONS:
Other: Virtual Reality application — Virtual Reality application with a VR goggle
  Arms: Virtual reality

SUMMARY:
This study is an experimental single centre study investigating the effect of VR on overall sleep quality and number of awakenings in patients with diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Able to speak Dutch/French
* Continuing usual care regarding medication use 3 weeks prior and during study participation
* Diagnosis of DPN for 6 months or longer, confirmed on EMG

Exclusion Criteria:

* History of seizures/epilepsia
* Susceptibility to motion sickness or cyber-sickness, susceptibility to claustrophobia
* shift workers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Change in sleep efficiency between experimental and control intervention. | Evaluated during two time periods of two weeks.
  Measured with actigraphy.
Change in number of awakenings during the night between experimental and control intervention. | Evaluated during two time periods of two weeks.
  Measured with actigraphy.

SECONDARY OUTCOMES:
Change in subjective sleep quality between experimental and control intervention. | Evaluated during two time periods of two weeks.
  Measured with the Pittsburgh Sleep Quality Index (ranging from 0-21 with higher scores a poorer sleep quality).
Change in pain intensity reporting between experimental and control intervention. | Evaluated during two time periods of two weeks.
  Measured with Visual Analogue Scale pain diary, whereby higher scores indicate hisger pain intensity.
Pain catastrophizing | Evaluated at the end of the experimental and control intervention namely after the two-week periods.
  Measured with the Pain Catastrophizing Scale whereby higher score are indicative for more catastrophizing.
Anxiety and depressive symptoms | Evaluated at the end of the experimental and control intervention namely after the two-week periods.
  Measured with the Hospital Anxiety and Depression Scale
Change in clinical status | Evaluated at the end of the experimental and control intervention namely after the two-week periods.
  Measured with the Global perceived effect
Any side effects of the experimental intervention | Evaluated at the end of the experimental intervention namely after the two-week period.
Nature, severity and impact of insomnia | Evaluated at the end of the experimental and control intervention namely after the two-week periods.
  Measured with the Insomnia Severity Index

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided